CLINICAL TRIAL: NCT02584634
Title: A PHASE 1B/2, OPEN-LABEL, DOSE-FINDING STUDY TO EVALUATE SAFETY, EFFICACY, PHARMACOKINETICS AND PHARMACODYNAMICS OF AVELUMAB (MSB0010718C) IN COMBINATION WITH EITHER CRIZOTINIB OR PF-06463922 IN PATIENTS WITH ADVANCED OR METASTATIC NON-SMALL CELL LUNG CANCER
Brief Title: Study to Evaluate Safety, Efficacy, Pharmacokinetics And Pharmacodynamics Of Avelumab In Combination With Either Crizotinib Or PF-06463922 In Patients With NSCLC. (Javelin Lung 101)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated since there was no need for further safety or efficacy data to be collected. The participants having benefit from the Investigational treatments have been moved to a continuation study (NCT05059522)
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B9991005; 2015-001879-43 (EudraCT Number); JAVELIN LUNG 101 (Other: Alias Study Number)
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Results first posted 2022-02-09 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; ALK; avelumab; crizotinib; PF-06463922
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — avelumab; lorlatinib; Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): ALK negative Non-Small Cell Lung Cancer
  Interventions: Drug: Avelumab; Drug: Crizotinib
- Group B (Experimental): ALK positive Non-Small Cell Lung Cancer
  Interventions: Drug: Avelumab; Drug: PF-06463922

INTERVENTIONS:
Drug: Avelumab — Administered by IV once every two weeks in doses of either 5 mg/kg or 10 mg/kg
  Other Names: MSB0010718C
Drug: PF-06463922 — Tablets taken orally once every day in doses of either 100mg, 75mg, or 50mg.
  Arms: Group B
Drug: Crizotinib — Capsules. Taken orally once or twice every day in doses of either 200mg or 250mg.
  Other Names: PF-02341066
  Arms: Group A

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of avelumab when combined with either crizotinib or PF-06463922.

DETAILED DESCRIPTION:
This is a Phase 1b/2, open label, multi center, multiple dose, safety, pharmacokinetic and pharmacodynamic study of Group A and Group B in cohorts of adult patients with locally advanced or metastatic NSCLC.

ELIGIBILITY:
* Inclusion Criteria
* Diagnosis of advanced or metastatic NSCLC. Group A must be ALK negative NSCLC and Group B must be ALK positive NSCLC
* Group A at least one prior regimen of therapy
* Group B any number of prior regimens.
* Mandatory tumor tissue available
* At least one measurable lesion
* ECOG Performance status 0 or 1
* Adequate bone marrow, renal, liver and pancreatic function
* Negative pregnancy test for females of childbearing potential
* Group B Phase 2: No prior systemic treatment for advanced or metastatic disease (adjuvant and/or neoadjuvant therapies are allowed if completed at least 6 months prior to study entry. No prior tyrosine kinase inhibitor therapy is allowed at any time prior to study entry)

Exclusion Criteria:

* No prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody.
* No Severe or Chronic medical conditions including gastrointestinal abnormalities or significant cardiac history
* No active infection requiring systemic therapy
* Prior organ transplantation including allogenic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2022-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (7):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ophthalmic Consultants of Boston Inc (OCB), Boston, Massachusetts
  - Tennessee Oncology, PLLC, Nashville, Tennessee
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Japan (3):
  - Aichi cancer center central hospital, Nagoya, Aichi-ken
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
- South Korea (3):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Institut Catala d'Oncologia de Badalona, Badalona, Barcelona
  - Hospital Quiron Barcelona, Barcelona
  - Hospital Universitari de la Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Solomon BJ, Dagogo-Jack I, Lee SH, Boyer MJ, Ramalingam SS, Carcereny E, Felip E, Han JY, Hida T, Hughes BGM, Kim SW, Nishio M, Seto T, Okamoto T, Zhang X, Martini JF, Wang E, De Beukelaer S, Bauer TM. Avelumab in Combination With Lorlatinib or Crizotinib in Patients With Previously Treated Advanced NSCLC: Phase 1b/2 Results From the JAVELIN Lung 101 Trial. JTO Clin Res Rep. 2024 May 16;5(7):100685. doi: 10.1016/j.jtocrr.2024.100685. eCollection 2024 Jul. PMID 39034968
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B9991005&StudyName=A%20Phase%201b%2F2%2C%20Open-label%2C%20Dose-finding%20Study%20To%20Evaluate%20Safety%2C%20Efficacy%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Avelumab%20%28msb0010718c%29%20In%20Combination%20With%20Either%20Crizotinib%20Or%20Pf-06463922%20In%20Patients%20With%20Advanced%20Or%20Metastatic%20Non-small%20Cell%20Lung%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Avelumab + Crizotinib: Participants with locally advanced or metastatic Anaplastic Lymphoma Kinase (ALK)-negative non-small cell lung cancer (NSCLC) received avelumab 10 mg/kg as a 1-hour intravenous (IV) infusion once every 2 weeks (Day 1 of each cycle) and crizotinib 250 mg (starting dose) orally twice a day (BID) on a continuous daily dosing schedule.
- Group B: Avelumab + Lorlatinib: Participants with locally advanced or metastatic ALK-positive NSCLC received avelumab 10 mg/kg as a 1-hour IV infusion once every 2 weeks (Day 1 of each cycle) and lorlatinib 100 mg (starting dose) orally once a day (QD) on a continuous daily dosing schedule.
Period: Overall Study
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Started | 12 | 31
Completed | 0 | 0
Not Completed | 12 | 31
Not completed — Adverse Event | 3 | 5
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Progressive disease | 7 | 15
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 0 | 6

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants who received at least one dose of study drug. Participants were classified according to the study treatment actually received. If a participant received more than one treatment the participant was classified according to the first treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib | Total
Number analyzed (Participants) | 12 | 31 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.67 (10.43) | 53.32 (11.59) | 54.81 (11.41)
Age, Customized [Number; unit: Participants]
  <65 years | 9 | 25 | 7
  65-<75 years | 2 | 5 | 2
  75-<85 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 19 | 25
  Male | 6 | 12 | 18
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 17 | 25
  White | 4 | 13 | 17
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 30 | 41
  Not Reported | 1 | 0 | 1
Age Range [Median (Full Range); unit: Years] | 59.5 [43 to 76] | 54 [30 to 77] | 55 [30 to 77]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs): Phase 1b
Description: Any of the following adverse events (AEs) occurring during the primary DLT observation period that are attributable to one, the other, or both study drugs were classified as DLTs: Grade 4 (life-threatening) neutropenia if >7 days in duration; febrile neutropenia; Grade >=3 (severe or life threatening) neutropenic infection; Grade >=3 thrombocytopenia with bleeding; Grade 4 thrombocytopenia >7 days; Grade 4 anemia; any Grade >=3 toxicity, except for any of the following: transient (<=6 hours) Grade 3 (severe) flu like symptoms or fever; transient (<=24 hours) Grade 3 fatigue, local reactions, or headache that resolved to Grade <=1 (no AE or mild AE); Grade 3 nausea and/or vomiting, diarrhea or skin toxicity that resolved to Grade <=1 within 7 days; any Grade >=3 amylase or lipase abnormality; tumor flare phenomenon; single laboratory values out of normal range that were not related to treatment, did not have any clinical correlate, and resolve to Grade <=1 within 7 days.
Time Frame: First 2 cycles (1 cycle = 14 days)
Population: The analysis population included all participants enrolled in Phase 1b who were in the safety analysis set (all participants who received at least one dose of study drug), and either experienced DLT during the first 2 cycles (1 cycle = 14 days), or completed the observation period for the first 2 cycles of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 12 | 28
Participants | 5 | 2

2. Primary Outcome: Percentage of Participants With Objective Response (OR): Phase 2
Description: OR is defined as complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 from start date (the date of first dose of study treatment) until disease progression or death due to any cause. Both CR and PR must be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response are first met. Per RECIST v1.1: CR is defined as the disappearance of all target or non-target lesions; any pathological lymph nodes (whether target or non target) must have reduction in short axis to <10 mm and all lymph nodes must be non-pathological in size (<10 mm short axis). PR is defined as a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Screening, Day 1 of each cycle starting Cycle 3, up to end of treatment/withdrawal (maximum of 5 years)
Population: The analysis population included all participants who received at least one dose of study drug. Participants were classified according to the study treatment actually received. If a participant received more than one treatment the participant was classified according to the first treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 12 | 31
Percentage of participants | 25.0 [5.5 to 57.2] | 51.6 [33.1 to 69.8]

3. Primary Outcome: Percentage of Participants With CR for Group B: Phase 2
Description: Per RECIST v1.1: CR is defined as the disappearance of all target or non-target lesions; any pathological lymph nodes (whether target or non target) must have reduction in short axis to <10 mm and all lymph nodes must be non-pathological in size (<10 mm short axis).
Time Frame: Baseline up to 60 months
Population: The analysis population included all participants who received at least one dose of study drug in Group B. Participants were classified according to the study treatment actually received. If a participant received more than one treatment the participant was classified according to the first treatment received. Results for Group A are not reported for this outcome measure according to the protocol.
Measure: Number; unit: Percentage of participants
Arm/Group | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 31
Percentage of participants | 3.2

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are those events with onset dates occurring during the on-treatment period for the first time, or if the worsening of an event is during the on-treatment period. Treatment-related AEs was any untoward medical occurrence attributed to study drug in a participant who received study drug. Per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03: Grade 3 (Severe) events=unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment; Grade 4 (Life-threatening) events caused participant to be in imminent danger of death; Grade 5 (Death) events=death related to an AE. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in participant hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to 30 days after last dose of study treatment or the day before start day of new anti-cancer therapy (maximum of 5 years)
Population: The analysis population included all participants who received at least one dose of study drug. Participants were classified according to the study treatment actually received. If a participant received more than one study treatment, the participant were classified according to the first treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 12 | 31
Participants
  Participants with TEAEs | 12 | 30
  Participants with Grade >= 3 TEAEs | 7 | 23
  Participants with treatment-related TEAEs | 12 | 28
  Participants with Grade >= 3 treatment-related TEAEs | 6 | 16
  Participants with SAEs | 5 | 21
  Participants with treatment-related SAEs | 2 | 6
  Participants with TEAEs leading to discontinuation of avelumab | 3 | 10
  Participants with TEAEs leading to discontinuation of crizotinib: number analyzed (Participants) | 12 | 0
  Participants with TEAEs leading to discontinuation of crizotinib | 6 |
  Participants with TEAEs leading to discontinuation of lorlatinib: number analyzed (Participants) | 0 | 31
  Participants with TEAEs leading to discontinuation of lorlatinib |  | 2
  Participants with TEAEs leading to discontinuation of any study drug | 6 | 10
  Participants with TEAEs leading to discontinuation of all study drugs | 3 | 1
  Participants with treatment-related TEAEs leading to discontinuation of avelumab | 2 | 9
  Participants with treatment-related TEAEs leading to discontinuation of crizotinib: number analyzed (Participants) | 12 | 0
  Participants with treatment-related TEAEs leading to discontinuation of crizotinib | 5 |
  Participants with treatment-related TEAEs leading to discontinuation of lorlatinib: number analyzed (Participants) | 0 | 31
  Participants with treatment-related TEAEs leading to discontinuation of lorlatinib |  | 2
  Participants with TEAEs leading to death | 1 | 4
  Participants with treatment-related TEAEs leading to death | 0 | 1
  Participants with infusion-related reactions | 5 | 9

5. Secondary Outcome: Number of Participants With Baseline Laboratory Abnormalities Grade <=2 and Post-Baseline Laboratory Abnormalities of Grades 3 or 4 Per NCI CTCAE v4.03
Description: The laboratory results were graded according to the NCI CTCAE v4.03 severity grade. Grade 1=mild AE. Grade 2=moderate AE. Grade 3=severe AE. Grade 4=life-threatening consequences; urgent intervention indicated. Shift tables were provided to examine the distribution of laboratory toxicities. The following parameters had met the criteria of CTCAE grade shift change from Grade <=2 at baseline to Grade 3 or 4 post baseline: anemia, lymphocyte count decreased, lymphocyte count decreased, neutrophil count decreased, white blood cell decreased, alanine aminotransferase increased, aspartate aminotransferase increased, blood bilirubin increased, cholesterol high, Creatine phosphokinase (CPK) increased, Gamma glutamyl transferase (GGT) increased, hypercalcemia, hyperglycemia, hypermagnesemia, hypertriglyceridemia, hypoalbuminemia, hyponatremia, lipase increased, serum amylase increased. Baseline is defined as the last assessment prior to the date/time of the first dose of study treatment.
Time Frame: Screening up to end of treatment/withdrawal (maximum of 5 years)
Population: The analysis population included all participants who received at least one dose of study drug and who could be evaluated for CTCAE criteria for each parameter in each treatment group. Participants were classified according to the study treatment actually received. If a participant received more than one study treatment, the participant was classified according to the first treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 12 | 31
Participants
  Anemia | 0 | 3
  Lymphocyte count decreased | 1 | 2
  Lymphocyte count increased | 0 | 2
  Neutrophil count decreased | 1 | 0
  White blood cell decreased | 1 | 0
  Alanine aminotransferase increased | 3 | 0
  Aspartate aminotransferase increased | 2 | 1
  Blood bilirubin increased | 0 | 1
  Cholesterol high | 0 | 5
  CPK increased: number analyzed (Participants) | 10 | 31
  CPK increased | 0 | 2
  GGT increased | 1 | 5
  Hypercalcemia | 0 | 2
  Hyperglycemia | 1 | 1
  Hypermagnesemia | 0 | 1
  Hypertriglyceridemia | 0 | 7
  Hypoalbuminemia | 0 | 1
  Hyponatremia | 1 | 3
  Lipase increased | 1 | 5
  Serum amylase increased | 0 | 1
  Hemoglobin increased | 0 | 0
  Platelet count decreased | 0 | 0
  Alkaline phosphatase increased | 0 | 0
  Creatinine increased | 0 | 0
  Hyperkalemia | 0 | 0
  Hypernatremia | 0 | 0
  Hypocalcemia | 0 | 0
  Hypoglycemia | 0 | 0
  Hypokalemia | 0 | 0
  Hypomagnesemia | 0 | 0
  Hypophosphatemia | 0 | 0

6. Secondary Outcome: Number of Participants With Vital Signs Meeting Pre-defined Criteria
Description: Pre-defined criteria in vital signs: pulse rate <50 beats per minute, pulse rate >120 bpm, sitting diastolic blood pressure (DBP) increase and decrease in change from baseline of >= 20 millimeter of mercury (mmHg), sitting systolic blood pressure(SBP) < 90 mmHg, increase and decrease in change from baseline of >= 30mmHg. Baseline is defined as the last assessment prior to the date/time of the first dose of study treatment.
Time Frame: Screening up to end of treatment/withdrawal (maximum of 5 years)
Population: The analysis population included all participants who received at least one dose of study drug. Participants were classified according to the study treatment actually received. If a participant received more than one study treatment, the participant was classified according to the first treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 12 | 31
Participants
  Pulse rate <50 bpm | 2 | 0
  Pulse rate >120 bpm | 0 | 4
  Sitting DBP change >= 20 mmHg increase | 2 | 13
  Sitting DBP change >= 20 mmHg decrease | 5 | 8
  Sitting SBP <90 mmHg | 1 | 4
  Sitting SBP change >= 30 mmHg increase | 1 | 11
  Sitting SBP change >= 30 mmHg decrease | 3 | 2

7. Secondary Outcome: Disease Control Rate (DCR)
Description: DC is defined as objective response (CR or PR) or stable disease (SD) per RECIST v.1.1 from the date of first dose of study treatment until disease progression or death due to any cause. The DCR is the proportion of patients with DC. Per RECIST v1.1: CR is defined as the disappearance of all target or non-target lesions; any pathological lymph nodes (whether target or non target) must have reduction in short axis to <10 mm. PR is defined as a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD is defined as a >=20% increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions.
Time Frame: Screening, Day 1 of each cycle starting Cycle 3, up to end of treatment/withdrawal (maximum of 5 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 12 | 31
Percentage of participants | 58.3 [27.7 to 84.8] | 71.0 [52.0 to 85.8]

8. Secondary Outcome: Duration of Response (DR)
Description: DR: time from first documented occurrence of response (PR or CR) until date of first documented PD or death due to underlying cancer. Per RECIST 1.1: CR: disappearance of all non-nodal target lesions and of all non-target lesions; any pathological lymph nodes assigned as target lesions/non-target lesions have a reduction in short axis to <10 mm. PR: at least a >=30% decrease in sum of diameter of all target lesions, taking as reference baseline sum of diameters. PD: at least a >=20% increase in sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. Appearance of new lesions. Participants with no PD and were still alive by 02 Feb 2020, were censored at last adequate tumor assessment. Kaplan-Meier method was used for DR analysis.
Time Frame: Screening, Day 1 of each cycle starting Cycle 3, up to end of treatment/withdrawal (maximum of 5 years)
Population: The analysis population included all participants who received at least one dose of study drug and who had confirmed complete response or partial response. Participants were classified according to the study treatment actually received. If a participant received more than one treatment the participant was classified according to the first treatment received.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 3 | 16
Month | 3.7 [3.7 to 4.6] | 14.7 [3.7 to NA] — The upper bound of the 95% confidence interval was not estimable due to limited number of events.

9. Secondary Outcome: Time to Tumor Response (TTR)
Description: TTR is defined, for participants with an objective response (CR or PR), as the time from the start date (the date of first dose of treatment) to the first documentation of objective response (CR or PR) which is subsequently confirmed. Per RECIST v1.1: CR: disappearance of all non-nodal target lesions and of all non-target lesions. In addition, any pathological lymph nodes assigned as target lesions/ non-target lesions must have a reduction in short axis to <10 mm. PR: at least a 30% decrease in sum of diameter of all target lesions, taking as reference baseline sum of diameters.
Time Frame: Screening, Day 1 of each cycle starting Cycle 3, up to end of treatment/withdrawal (maximum of 5 years)
Population: as for outcome 8
Measure: Median (Full Range); unit: Months
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 3 | 16
Months | 1.4 [1.4 to 6.9] | 1.8 [1.3 to 3.7]

10. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from start date (the date of first dose of treatment) to the date of the first documentation of PD per RECIST v1.1 or death due to any cause, whichever occurs first. Per RECIST v1.1: PD: a >=20% increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Screening, Day 1 of each cycle starting Cycle 3, up to end of treatment/withdrawal (maximum of 5 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 12 | 31
Months | 3.7 [1.5 to 5.5] | 6.4 [3.7 to 9.2]

11. Secondary Outcome: Kaplan-Meier Estimates of Overall Survival (OS)
Description: OS is defined as the time from start date (the date of first dose of treatment) to the date of death due to any cause.
Time Frame: Screening, Day 1 of each cycle starting Cycle 3, up to end of treatment/withdrawal (maximum of 5 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 12 | 31
Months | 16.4 [5.4 to 27.6] | 32.9 [10.7 to NA] — The upper bound of the 95% confidence interval was not estimable due to limited number of events.

12. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Crizotinib in The Presence of Avelumab
Description: Cmax of crizotinib in the presence of avelumab was observed directly from data.
Time Frame: Pre-dose, 1, 2, 4, 6 and 8 hours post dose on Day 1 of Cycle 2
Population: The analysis population included participants who received at least one dose of study drug and who had at least one of the pharmacokinetic (PK) parameters of interest for crizotinib in Group A. Group B was not evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Group A: Avelumab + Crizotinib
Number analyzed (Participants) | 10
nanograms per millilitre (ng/mL) | 281 (74)

13. Secondary Outcome: Time to Cmax (Tmax) of Crizotinib in The Presence of Avelumab
Description: Tmax of crizotinib in the presence of avelumab was observed directly from data as time of first occurrence.
Time Frame: Pre-dose, 1, 2, 4, 6 and 8 hours post dose on Day 1 of Cycle 2
Population: The analysis population included participants who received at least one dose of study drug and who had at least one of the PK parameters of interest for crizotinib in Group A. Group B was not evaluable for this outcome measure.
Measure: Median (Full Range); unit: Hours
Arm/Group | Group A: Avelumab + Crizotinib
Number analyzed (Participants) | 10
Hours | 2.03 [0.00 to 8.08]

14. Secondary Outcome: Area Under The Plasma Concentration-Time Curve During The Dosing Interval Time Course (AUCtau) of Crizotinib in The Presence of Avelumab
Description: AUCtau of crizotinib in the presence of avelumab was calculated by Linear/Log trapezoidal method. Dose interval is defined as after single dose from time zero to the next dose (after single dose and at steady state).
Time Frame: Pre-dose, 1, 2, 4, 6 and 8 hours post dose on Day 1 of Cycle 2
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per millilitre (ng*h/mL)
Arm/Group | Group A: Avelumab + Crizotinib
Number analyzed (Participants) | 10
nanograms*hours per millilitre (ng*h/mL) | 2755 (82)

15. Secondary Outcome: Apparent Plasma Clearance (CL/F) of Crizotinib in The Presence of Avelumab
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Pre-dose, 1, 2, 4, 6 and 8 hours post dose on Day 1 of Cycle 2
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Group A: Avelumab + Crizotinib
Number analyzed (Participants) | 10
Liter per hour (L/h) | 90.76 (82)

16. Secondary Outcome: Cmax of Crizotinib Metabolite PF-06260182 in The Presence of Avelumab
Description: Cmax of crizotinib metabolite PF-06260182 in the presence of avelumab was observed directly from data.
Time Frame: Pre-dose, 1, 2, 4, 6 and 8 hours post dose on Day 1 of Cycle 2
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group A: Avelumab + Crizotinib
Number analyzed (Participants) | 10
ng/mL | 84.11 (91)

17. Secondary Outcome: Tmax of Crizotinib Metabolite PF-06260182 in The Presence of Avelumab
Description: Tmax of crizotinib metabolite PF-06260182 in the presence of avelumab was observed directly from data as time of first occurrence.
Time Frame: Pre-dose, 1, 2, 4, 6 and 8 hours post dose on Day 1 of Cycle 2
Population: as for outcome 13
Measure: Median (Full Range); unit: Hours
Arm/Group | Group A: Avelumab + Crizotinib
Number analyzed (Participants) | 10
Hours | 3.02 [0.00 to 8.08]

18. Secondary Outcome: AUCtau of Crizotinib Metabolite PF-06260182 in The Presence of Avelumab
Description: AUCtau of crizotinib metabolite PF-06260182 in the presence of avelumab was calculated by Linear/Log trapezoidal method. Dose interval: single dose from time zero to the next dose (after single dose and at steady state).
Time Frame: Pre-dose, 1, 2, 4, 6 and 8 hours post dose on Day 1 of Cycle 2
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group A: Avelumab + Crizotinib
Number analyzed (Participants) | 10
ng*h/mL | 789.1 (116)

19. Secondary Outcome: Metabolite to Parent Ratio for AUCtau (MRAUCtau) of PF-06260182 in The Presence of Avelumab
Description: MRAUCtau of metabolite PF-06260182 in the presence of avelumab was calculated (MRAUCtau=Metabolite AUCtau/parent AUCtau). Parent=crizotinib, metabolite=PF-06260182
Time Frame: Pre-dose, 1, 2, 4, 6 and 8 hours post dose on Day 1 of Cycle 2
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Group A: Avelumab + Crizotinib
Number analyzed (Participants) | 10
Ratio | 0.2779 (33)

20. Secondary Outcome: Metabolite to Parent Ratio for Cmax (MRCmax) of PF-06260182 in The Presence of Avelumab
Description: MRCmax of metabolite PF-06260182 in the presence of avelumab was calculated (MRCmax=Metabolite Cmax/parent Cmax). Parent=crizotinib, metabolite=PF-06260182
Time Frame: Pre-dose, 1, 2, 4, 6 and 8 hours post dose on Day 1 of Cycle 2
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Group A: Avelumab + Crizotinib
Number analyzed (Participants) | 10
Ratio | 0.2902 (25)

21. Secondary Outcome: Cmax of Lorlatinib in The Presence of Avelumab
Description: Cmax of lorlatinib in the presence of avelumab was observed directly from data.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, and 24 hours (prior to Day 2 lorlatinib dose) post dose on Day 1 of Cycle 2
Population: The analysis population included participants who received at least one dose of study drug and who had at least one of the PK parameters of interest for lorlatinib in Group B. Group A is not evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 26
ng/mL | 596.9 (33)

22. Secondary Outcome: Tmax of Lorlatinib in The Presence of Avelumab
Description: Tmax of lorlatinib in the presence of avelumab was observed directly from data.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, and 24 hours (prior to Day 2 lorlatinib dose) post dose on Day 1 of Cycle 2
Population: as for outcome 21
Measure: Median (Full Range); unit: Hours
Arm/Group | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 26
Hours | 1.23 [0.933 to 4.33]

23. Secondary Outcome: AUCtau of Lorlatinib in The Presence of Avelumab
Description: AUCtau of lorlatinib in the presence of avelumab was calculated by Linear/Log trapezoidal method. Dose interval: single dose from time zero to the next dose (after single dose and at steady state).
Time Frame: Pre-dose, 1, 2, 4, 6, 8, and 24 hours (prior to Day 2 lorlatinib dose) post dose on Day 1 of Cycle 2
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 19
ng*h/mL | 5807 (42)

24. Secondary Outcome: Area Under The Plasma Concentration Time Curve From Time of Dosing to The Last Collection Time Point (AUClast) of Lorlatinib in The Presence of Avelumab
Description: AUClast of lorlatinib in the presence of avelumab.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, and 24 hours (prior to Day 2 lorlatinib dose) post dose on Day 1 of Cycle 2
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 26
ng*h/mL | 4872 (52)

25. Secondary Outcome: CL/F of Lorlatinib in The Presence of Avelumab
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, and 24 hours (prior to Day 2 lorlatinib dose) post dose on Day 1 of Cycle 2
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 19
L/h | 16.97 (44)

26. Secondary Outcome: Cmax of Avelumab in The Presence of Crizotinib (Group A) or Lorlatinib (Group B) After Single Dose of Avelumab
Description: Cmax of avelumab in the presence of crizotinib was observed directly from the data in Group A. Cmax of avelumab in the presence of lorlatinib was observed directly from the data in Group B.
Time Frame: Pre-dose, 1, and 168 hours post dose of avelumab on Cycle 1 Day 1.
Population: The analysis population included participants who received at least one dose of study drug and who had at least one post-dose concentration measurement above the lower limit of quantification for avelumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (ug/mL)
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 8 | 16
micrograms/milliliter (ug/mL) | 193.2 (14) | 195.7 (28)

27. Secondary Outcome: Cmax of Avelumab in The Presence of Crizotinib (Group A) or Lorlatinib (Group B) After Multiple Doses of Avelumab
Description: as for outcome 26
Time Frame: Pre-dose, 1, and 168 hours post dose of avelumab on Cycle 2 Day 1
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 8 | 17
ug/mL | 174.5 (35) | 169.4 (68)

28. Secondary Outcome: Trough Serum Concentration (Ctrough) of Avelumab in The Presence of Crizotinib (Group A) Following Multiple Doses of Avelumab
Description: Ctrough is defined as predose concentration following multiple doses. Ctrough of avelumab in the presence of crizotinib was observed directly from the data in Group A.
Time Frame: Pre-dose on Day 1 of Cycles 2-5, 11, 17, 23, 29, 35, and 47.
Population: The analysis population included participants who received at least one dose of study drug and who had least one observation. Number of Participants Analyzed represents the total number of participants in the analysis population for this outcome measure. Number Analyzed represents the number of participants with concentration measurement above lower limit of quantification at each visit. Group B was not evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Group A: Avelumab + Crizotinib
Number analyzed (Participants) | 12
ug/mL
  Cycle 2 Day 1: number analyzed (Participants) | 7
  Cycle 2 Day 1 | 11.76 (68)
  Cycle 3 Day 1: number analyzed (Participants) | 6
  Cycle 3 Day 1 | 16.26 (53)
  Cycle 4 Day 1: number analyzed (Participants) | 7
  Cycle 4 Day 1 | 16.71 (34)
  Cycle 5 Day 1: number analyzed (Participants) | 5
  Cycle 5 Day 1 | 14.21 (46)
  Cycle 11 Day 1: number analyzed (Participants) | 2
  Cycle 11 Day 1 | 26.64 (4)
  Cycle 17 Day 1: number analyzed (Participants) | 2
  Cycle 17 Day 1 | 30.59 (9)
  Cycle 23 Day 1: number analyzed (Participants) | 2
  Cycle 23 Day 1 | 30.63 (15)
  Cycle 29 Day 1: number analyzed (Participants) | 2
  Cycle 29 Day 1 | 30.72 (55)
  Cycle 35 Day 1: number analyzed (Participants) | 2
  Cycle 35 Day 1 | 37.31 (27)
  Cycle 47 Day 1: number analyzed (Participants) | 2
  Cycle 47 Day 1 | 40.91 (15)

29. Secondary Outcome: Trough Serum Concentration (Ctrough) of Avelumab in The Presence of Lorlatinib (Group B) Following Multiple Doses of Avelumab
Description: Ctrough is defined as predose concentration following multiple doses. Ctrough of avelumab in the presence of lorlatinib was observed directly from the data in Group B.
Time Frame: Pre-dose on Day 1 of Cycles 2-5, 11, 17, 23, 29, 35, 41, and 47.
Population: The analysis population included participants who received at least one dose of study drug and who had least one observation. Number of Participants Analyzed represents the total number of participants in the analysis population for this outcome measure. Number Analyzed represents the number of participants with concentration measurement above lower limit of quantification at each visit. Group A was not evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 25
ug/mL
  Cycle 2 Day 1: number analyzed (Participants) | 22
  Cycle 2 Day 1 | 16.86 (88)
  Cycle 3 Day 1: number analyzed (Participants) | 19
  Cycle 3 Day 1 | 16.99 (116)
  Cycle 4 Day 1: number analyzed (Participants) | 21
  Cycle 4 Day 1 | 23.71 (80)
  Cycle 5 Day 1: number analyzed (Participants) | 16
  Cycle 5 Day 1 | 26.74 (68)
  Cycle 11 Day 1: number analyzed (Participants) | 15
  Cycle 11 Day 1 | 31.31 (71)
  Cycle 17 Day 1: number analyzed (Participants) | 13
  Cycle 17 Day 1 | 32.69 (60)
  Cycle 23 Day 1: number analyzed (Participants) | 11
  Cycle 23 Day 1 | 33.20 (56)
  Cycle 29 Day 1: number analyzed (Participants) | 10
  Cycle 29 Day 1 | 25.77 (66)
  Cycle 35 Day 1: number analyzed (Participants) | 10
  Cycle 35 Day 1 | 31.27 (47)
  Cycle 41 Day 1: number analyzed (Participants) | 7
  Cycle 41 Day 1 | 30.81 (59)
  Cycle 47 Day 1: number analyzed (Participants) | 8
  Cycle 47 Day 1 | 39.63 (64)

30. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) Against Avelumab by Never and Ever Positive Status
Description: ADA never-positive was defined as no positive ADA results at any time point. ADA ever-positive was defined as at least one positive ADA result at any time point. Baseline is defined as the last assessment on or prior to the date/time of the first dose of avelumab.
Time Frame: Day 1 of Cycles 1-5, then every 12 weeks thereafter, end of treatment/withdrawal, and 30 days after last avelumab dose (up to a maximum of 5 years)
Population: The analysis population was a subset of the safety analysis set (all participants who received at least one dose of study drug) and included participants who had at least one ADA sample collected for avelumab.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Including all the participants from Group A and Group B.
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib | All Participants
Number analyzed (Participants) | 12 | 31 | 43
Participants
  ADA never-positive | 9 | 25 | 34
  ADA ever-positive | 3 | 6 | 9

31. Secondary Outcome: Number of Participants With Positive Programmed Death Ligand-1 (PD-L1) Biomarker Expression
Description: PD-L1 protein expression is determined by using Combined Positive Score (CPS), which is the percentage of viable tumor and tumor-infiltrated immune cells (restricted to lymphocytes and macrophages) within or directly associated with tumor cell strands showing partial or complete membrane staining using the SP263 antibody. Positive is defined as CPS>=1% and negative is defined as CPS <1%.
Time Frame: Baseline
Population: The analysis population was a subset of the safety analysis set (all participants who received at least one dose of study drug) and included participants who had at least one biomarker parameter of PD-L1 from the corresponding assay sample with at least one baseline biomarker measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 9 | 24
Participants
  Positive | 7 | 20
  Negative | 2 | 4

32. Secondary Outcome: Number of Participants With Positive Tumor Infiltrating CD8+ Lymphocytes
Description: Tumor infiltrating CD8+ lymphocytes is defined as the number of CD8+ cells per unit area and the percent of counted cells. Positive is defined as >=1% and negative is defined as <1%.
Time Frame: Baseline
Population: The analysis population was a subset of the safety analysis set (all participants who received at least one dose of study drug) and included participants who had at least one biomarker parameter of tumor infiltrating CD8+ lymphocytes from the corresponding assay sample with at least one baseline biomarker measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
Number analyzed (Participants) | 10 | 22
Participants
  Positive | 6 | 4
  Negative | 4 | 18

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days post lost dose of study treatment with a maximum of 5 years
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Group A: Avelumab + Crizotinib | Group B: Avelumab + Lorlatinib
All-Cause Mortality (participants affected / at risk) | 10/12 | 15/31
Serious Adverse Events (participants affected / at risk) | 5/12 | 21/31
Other Adverse Events (participants affected / at risk) | 12/12 | 28/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Avelumab + Crizotinib (N=12) | Group B: Avelumab + Lorlatinib (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Disease progression (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
Postoperative wound infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system vasculitis (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2
Delirium (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Superior vena cava occlusion (Vascular disorders) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sudden death (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Avelumab + Crizotinib (N=12) | Group B: Avelumab + Lorlatinib (N=31)
Anaemia (Blood and lymphatic system disorders) | 3 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 2
Pericardial effusion (Cardiac disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 8
Dry eye (Eye disorders) | 1 | 1
Keratitis (Eye disorders) | 1 | 0
Asthenia (General disorders) | 2 | 3
Chest pain (General disorders) | 0 | 4
Chills (General disorders) | 3 | 2
Fatigue (General disorders) | 1 | 4
Hypothermia (General disorders) | 1 | 0
Localised oedema (General disorders) | 0 | 2
Mucosal inflammation (General disorders) | 2 | 0
Oedema (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 12
Peripheral swelling (General disorders) | 0 | 2
Pyrexia (General disorders) | 3 | 5
Swelling face (General disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 7
Dry mouth (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 7 | 5
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 6 | 6
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 3
Conjunctivitis (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 3
Rhinitis (Infections and infestations) | 0 | 2
Tooth abscess (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 5
Urinary tract infection (Infections and infestations) | 0 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 6
Procedural pain (Injury, poisoning and procedural complications) | 1 | 2
Alanine aminotransferase increased (Investigations) | 4 | 9
Amylase increased (Investigations) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 7
Blood alkaline phosphatase increased (Investigations) | 1 | 2
Blood cholesterol increased (Investigations) | 0 | 19
Blood creatine phosphokinase increased (Investigations) | 1 | 4
Blood creatinine increased (Investigations) | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 3
Hypophonesis (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 5
Neutrophil count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 0 | 8
White blood cell count decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 18
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Carpal tunnel syndrome (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 4
Dysgeusia (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 4
Hemiparesis (Nervous system disorders) | 1 | 1
Lethargy (Nervous system disorders) | 0 | 3
Memory impairment (Nervous system disorders) | 0 | 3
Migraine (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 7
Paraesthesia (Nervous system disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 5
Somnolence (Nervous system disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 2
Hallucination, visual (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 6
Haematuria (Renal and urinary disorders) | 0 | 2
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 3
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 5
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2
Blood triglycerides increased (Investigations) | 0 | 2
Hyperaesthesia (Nervous system disorders) | 0 | 2
Restlessness (Psychiatric disorders) | 0 | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Enrollment in the study was terminated early based on the changing landscape in treatment options for treatment naïve ALK positive NSCLC. This decision was not due to any safety concerns or regulatory interactions. All participants on active treatment at the time of the early enrollment termination could continue treatment and follow up per the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT02584634/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT02584634/SAP_001.pdf